CLINICAL TRIAL: NCT01383278
Title: Evaluation of a Computer-Delivered 5 A's Intervention for Smoking
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient sample size to complete study and merged with parent grant funded study
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: SBIRTCSVCU; R01DA026091 (NIH)
Record Dates: First submitted 2011-06-24; First posted 2011-06-28 (Estimated); Last update posted 2015-12-21 (Estimated); Status verified 2015-12

CONDITIONS: Smoking
Keywords: tobacco; smoking; smoking cessation
MeSH Terms: conditions — Smoking; Smoking Cessation | interventions — Smoking Devices; Mass Screening

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Computer-directed 5 A's intervention for smoking (Experimental)
  Interventions: Behavioral: Computer-directed 5 A's intervention for smoking
- Screening and resource provision (Active Comparator)
  Interventions: Behavioral: Screening and resource provision

INTERVENTIONS:
Behavioral: Computer-directed 5 A's intervention for smoking — Computer-directed 5 A's intervention for smoking
  Arms: Computer-directed 5 A's intervention for smoking
Behavioral: Screening and resource provision — Screening and resource provision
  Arms: Screening and resource provision

SUMMARY:
This is a 2-group RCT in 380 tobacco-using medical patients that will compare a single session, computer-directed 5 A's intervention for smoking (experimental condition) to screening and resource provision (control condition). Follow-up visits will occur at 1 and 3 months post study enrollment. Measures will focus on tobacco use and related psychosocial outcomes (e.g. mood, stress). We will compare resources used and economic costs needed to implement each intervention.

The Investigators hypothesize that patients receiving the computer-directed intervention will have significantly higher tobacco abstinence rates at 3 months post study enrollment compared to the control group. If indeed the computerized intervention increases tobacco abstinence rates compared to the control group, this intervention could be used to increase access to treatment for the millions of US smokers, ultimately reducing tobacco mortality and morbidity rates in this country.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 65 years
* Primary care patient
* Smoked at least one cigarette per day for the past seven days or at least 10 cigarettes total during the past week
* Smoked at least 100 cigarettes (lifetime)
* Had no recent (past 90 days) use of other forms of tobacco (pipes, cigars, NRT)
* Able to speak English

Exclusion Criteria:

- Pregnant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2012-02; Primary Completion 2012-09 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Tobacco use | 3 months post-randomization
  The primary outcome variable for this study will be smoking cessation at 3 month follow-up as measured by self-report, salivary cotinine and carbon monoxide levels.

SECONDARY OUTCOMES:
Mood and stress | 3 months post-randomization
  By using the K-10 Instrument
Resource utilization and economic costs | 3 months post-randomization

CONTACTS AND LOCATIONS:
Overall Officials: Dace Svikis, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States